CLINICAL TRIAL: NCT06931834
Title: Expanded Access Treatment Protocol for R007 (Probucol) Tablets in Adults With Genetically-Confirmed Mitochondrial Disease and Chronic Kidney Disease (Intermediate-Size Patient Population)
Brief Title: Expanded Access Program for R007 (Probucol) Tablets in Adults With Mitochondrial Disease and Chronic Kidney Disease
Status: Available | Type: Expanded Access
Sponsor: RiboNova Inc. (Industry)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: EP2025010101
Record Dates: First submitted 2025-04-04; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Mitochondrial Disease; Chronic Kidney Disease
Keywords: Mitochondrial disease; Chronic kidney disease; Myopathy; Genetic disease; Rare disease; Probucol
MeSH Terms: conditions — Mitochondrial Diseases; Renal Insufficiency, Chronic; Muscular Diseases; Genetic Diseases, Inborn; Rare Diseases | interventions — Probucol

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Probucol — Probucol 250 mg tablets orally up to a daily dose of 1,000 mg
  Other Names: R007; Lorelco

SUMMARY:
The purpose of this expanded access program is to enable access to R007 (probucol) tablets for the compassionate treatment of adults with mitochondrial disease who also have chronic kidney disease.

DETAILED DESCRIPTION:
The protocol for this expanded access program provides for the compassionate treatment with R007 (probucol) tablets of adults who (i) have serious or life-threatening mitochondrial disease and also have chronic kidney disease stages 3 or 4, (ii) do not have access to a satisfactory alternative therapy to treat their condition, and (iii) are not able to enroll in a clinical trial.

ELIGIBILITY:
Inclusion Criteria

A patient must meet all of the following criteria to be eligible:

1. Age 18 to 75 years inclusive;
2. Diagnosis of genetically-confirmed mitochondrial disease with a pathogenic mutation or defect in their mitochondrial or nuclear DNA;
3. Diagnosis of chronic kidney disease stage 3 or stage 4;
4. Moderate or severe symptomatology of mitochondrial disease;
5. A sexually-active patient agrees to practice acceptable methods of contraception throughout the protocol period;
6. The patient is not eligible for, or does not have access to, a clinical trial;
7. The patient (or guardian/legal representative) provides signed and dated informed consent to be treated with probucol in accordance with the expanded access protocol.

Exclusion Criteria

A patient who meets any of the following criteria will not be eligible:

1. A known hypersensitivity or adverse reaction to probucol;
2. A medical condition or laboratory result that, in the opinion of the treating physician, will interfere with the safe completion of the protocol;
3. An active fungal infection, acute blood, lung, or bladder infection, clinically significant hepatic or renal dysfunction, and/or viral infection (past or present) that, in the opinion of the treating physician, may have a clinically significant effect on their treatment;
4. Taking an investigational drug other than probucol within one month prior to the first dosing with probucol under the protocol;
5. A medical history or condition that increases the potential for QTc prolongation;
6. A female with a positive pregnancy test result or who is breastfeeding;
7. Has received or is receiving kidney dialysis;
8. Has received or is scheduled to receive an organ transplant;
9. Known or suspected active alcohol and/or substance abuse;
10. A history of or current suicidal ideation, behavior, and/or attempts; or
11. Is unable to swallow tablets or requires gastric feeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Zarazuela Zolkipli-Cunningham, MBChB, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States